CLINICAL TRIAL: NCT03980080
Title: Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation Study for the Assessment of Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of Single and Multiple Ascending Intravenous and Subcutaneous Doses of OSE-127 in Healthy Subjects
Brief Title: Phase I Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of OSE-127 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OSE Immunotherapeutics (Industry)
Collaborators: Servier (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OSE-127-C101; 2018-001832-22 (EudraCT Number)
Record Dates: First submitted 2019-05-13; First posted 2019-06-10 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Healthy Subjects
Keywords: CD127/IL-7Rα Antagonist; Auto-Immune Diseases; inflammatory bowel diseases; Ulcerative Colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: Part 1 (SAD) primary objective : safety and tolerability profile of single ascending IV (Cohort A) and SC (Cohort B) doses given to healthy subjects, compared to placebo.
  Part 2 (MAD) primary objective : safety and tolerability profile of two IV doses given on two separate occasions to healthy subjects, compared to placebo.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- OSE-127: Part 1 (SAD), Cohort A & Cohort B (Experimental)
  Interventions: Drug: OSE-127
- Placebo: Part 1 (SAD), Cohort A & Cohort B (Placebo Comparator)
  Interventions: Drug: Placebo
- OSE-127: Part 2 (MAD) (Experimental)
  Interventions: Drug: OSE-127
- Placebo: Part 2 (MAD) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OSE-127 — mAb antagonist to CD127 receptor (or IL-7Rα)
  Group 1-7
  6 escalating dose level groups IV
  SC
  Arms: OSE-127: Part 1 (SAD), Cohort A & Cohort B
Drug: Placebo — Vehicle study drug
  Arms: Placebo: Part 1 (SAD), Cohort A & Cohort B; Placebo: Part 2 (MAD)
Drug: OSE-127 — mAb antagonist to CD127 receptor (or IL-7Rα)
  Group 8-9
  2 escalating dose level groups IV
  Arms: OSE-127: Part 2 (MAD)

SUMMARY:
This study is a first-in-human phase I randomised, double-blind, placebo-controlled, evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of Single (IV and SC) and Multiple (IV only) Ascending Doses of OSE-127 in Healthy Subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18 to 65 years (extremes included). Maximum two subjects aged between 60 and 65 (extremes included) are allowed per dose group.
2. Healthy volunteers (medically stable), as determined on the basis of medical history, vital signs, clinical laboratory testing, and general physical examination performed at screening and deemed appropriate by the Investigator.
3. Electrocardiogram (ECG) within normal range, or showing no clinically relevant deviations, as judged by the Investigator.
4. Weighs at least 50 kg and no more than 100 kg and has a Body Mass Index (BMI) within normal range: 19.0 ≤ BMI ≤ 30.0 kg/m².
5. Negative urine test for selected drugs of abuse at screening.
6. Negative alcohol breath test at screening.
7. Female subjects is postmenopausal, surgically sterile (having had a hysterectomy or bilateral oophorectomy) and/or is using a highly effective method of contraception (from 2 weeks before first study drug administration until 28 days after the last follow-up visit, when it is confirmed that the RO of the subject <20% or 5 t1/2 whichever is longer).
8. Female subject has a negative pregnancy test at screening.
9. Non-vasectomized male subjects having a female partner of childbearing potential must agree to the use of a highly effective method of contraception (from the first study drug administration until 28 days after the last follow-up visit, when it is confirmed that the RO of the subject <20% or 5 t1/2 whichever is longer).
10. Willing to adhere to the prohibitions and restrictions specified in the protocol.
11. Informed Consent Form (ICF) signed voluntarily before any study-related procedure is performed, indicating that the subject understands the purpose of and procedures required for the study and is willing to participate in the study.
12. Non-smoker or light smoker, i.e. smokes maximal 5 cigarettes (or 3 cigars or 3 pipe-full) per day, and ability and willingness to refrain from smoking during confinement and ambulant visits in the CPU.

Exclusion Criteria:

1. A history of any clinically significant (as determined by the Investigator) cardiac, endocrinology, hematology, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other major disease or malignancy excluding non-melanoma skin cancer.
2. A known allergy, hypersensitivity, or intolerance to any of the excipients in the formulation of the study drug.
3. The subject has a history of severe allergic or anaphylactic reactions.
4. The suject has a history of consuming more than 14 units of alcoholic beverages per week for male subjects, and more than 10 units for females. Or a history of alcoholism, or drug/chemical/substance abuse within the past 2 years prior to screening.
5. Evidence or history of any clinically significant infections within the past 3 months.
6. Subject with known clinically relevant immunological disorders, or auto-immune disorders (e.g. rheumatoid arthritis, lupus erythematosus, scleroderma, etc...).
7. A positive hepatitis panel (including hepatitis B surface antigen [HBsAg] and anti-hepatitis C virus [HCV] antibodies [Abs]) or positive human immunodeficiency virus (HIV) antibody screens.
8. The subject has a supine systolic blood pressure (SBP) <90 or >149 mmHg and/or a diastolic blood pressure (DBP) <45 or >90 mmHg, and/or a pulse rate higher than 100 beats per minute (bpm) at screening (blood pressure measurements taken after subject has been resting in a supine position for a minimum of 5 minutes).
9. Pregnant or breastfeeding women.
10. The subject has received a live vaccine (excluding flu vaccination), within 30 days prior to study drug administration, or plan to receive this type of vaccine during the study.
11. The subject has received any systemic immunosuppressant agent, within 6 months prior to study drug administration.
12. The subject has received any antibody or biologic medicinal product, within 6 months prior to study drug administration.
13. The subject has received any systemic steroid, within 2 months prior to study drug administration.
14. Use of a prohibited therapy during the study.
15. Receipt of any investigational drug, within 30 days or 5 half-lives (whichever is longer) prior to the initial study drug administration.
16. The subject is participating in another clinical trial or has participated in another dose group of the current trial. Participation in non-interventional registries or epidemiological studies is allowed.
17. Having had a significant blood loss (including blood donation [>500 mL]) or a having had a transfusion of any blood product (within the past 60 days) or donated plasma (within 7 days prior to the initial study drug administration).
18. A condition that, in the opinion of the Investigator, could compromise their well-being or the course of the study, or prevent them from meeting or performing any study requirement.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2019-11-04 (Actual)

PRIMARY OUTCOMES:
Part 1 (SAD) & Part 2 (MAD) : Number of Participants With Treatment Emergent Adverse Events (TEAEs) | 12 weeks (for Part 1); 19 weeks (for Part 2)
Part 1 (SAD) & Part 2 (MAD) : Number of Participants With Clinically Significant Findings in Physical Examinations Reported as Adverse Event | 12 weeks (for Part 1); 19 weeks (for Part 2)
Part 1 (SAD) & Part 2 (MAD) : Number of Participants With Clinically Significant Change in Clinical Laboratory Results Reported as Adverse Event | 12 weeks (for Part 1); 19 weeks (for Part 2)
Part 1 (SAD) & Part 2 (MAD) :Number of Participants With Clinically Significant Change in Electrocardiogram (ECG) Reported as Adverse Event | 12 weeks (for Part 1); 19 weeks (for Part 2)
Part 1 (SAD) & Part 2 (MAD) :Number of Participants With Clinically Significant Change in vital signs Reported as Adverse Event | 12 weeks (for Part 1); 19 weeks (for Part 2)
Part 1 (SAD) & Part 2 (MAD) :Number of Participants With Clinically Significant Findings in Telemetry Reported as Adverse Event | 12 weeks (for Part 1); 19 weeks (for Part 2)
Part 1 (SAD) & Part 2 (MAD) : Incidence of anti-drug antibody (ADA) formation | 12 weeks (for Part 1); 19 weeks (for Part 2)

SECONDARY OUTCOMES:
Part 1 (SAD) & Part 2 (MAD) : Maximum Plasma Concentration [Cmax] | 12 weeks (for Part 1); 19 weeks (for Part 2)
Part 1 (SAD) & Part 2 (MAD) : Average serum Concentration over the dosing interval [Cavg] | 12 weeks (for Part 1); 19 weeks (for Part 2)
Part 1 (SAD) & Part 2 (MAD) : Trough serum Concentration observed at the end of the dosing interval [Ctrough] | 12 weeks (for Part 1); 19 weeks (for Part 2)
Part 1 (SAD) & Part 2 (MAD) : Elimination half-life associated with the terminal rate constant (λz) [T1/2] | 12 weeks (for Part 1); 19 weeks (for Part 2)
Part 1 (SAD) & Part 2 (MAD) : Time corresponding to the Cmax [Tmax] | 12 weeks (for Part 1); 19 weeks (for Part 2)
Part 1 (SAD) & Part 2 (MAD) : Area Under the serum concentration-time Curve from time zero till X days postdose [AUCτ] | 12 weeks (for Part 1); 19 weeks (for Part 2)
Part 1 (SAD) & Part 2 (MAD) : AUC calculated between time of administration and last quantifiable concentration [AUClast] | 12 weeks (for Part 1); 19 weeks (for Part 2)
Part 1 (SAD) & Part 2 (MAD) : AUC extrapolated to infinity [AUCinf] | 12 weeks (for Part 1); 19 weeks (for Part 2)
Part 1 (SAD) & Part 2 (MAD) : AUC over the dosing interval [AUC0-τ]. | 12 weeks (for Part 1); 19 weeks (for Part 2)
Part 1 (SAD) & Part 2 (MAD) : Accumulation Ratio [Rac]. | 12 weeks (for Part 1); 19 weeks (for Part 2)
Part 1 (SAD) & Part 2 (MAD) : CD-127 Receptor Occupancy [RO] | 12 weeks (for Part 1); 19 weeks (for Part 2)
Part 1 (SAD) & Part 2 (MAD) : Effect on total lymphocyte count | 12 weeks (for Part 1); 19 weeks (for Part 2)

CONTACTS AND LOCATIONS:
Overall Officials: Frédérique Corallo, MD, Study Director — OSE Immunotherapeutics
Locations (1):
- SGS Life Sciences (SGS LS), Clinical Pharmacology Unit (CPU), Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided